CLINICAL TRIAL: NCT01537796
Title: Comparison of a Technology-based System and an In-person Behavioral Weight Loss Intervention in the Severely Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO11120127
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Obesity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- In-Person weight loss (Experimental): Participants will attend weekly group intervention meetings. These sessions will address barriers associated with altering physical activity participation and dietary intake. Group discussions will be facilitated by the interventionist and interactive participation will be encouraged. Participants will be provided with written materials at each meeting to supplement group discussions. Paper diaries will be provided each week to assist participants with self-monitoring of calorie and fat consumption, and physical activity minutes and intensity. Participants will return the diary to the intervention staff each week for review and constructive feedback.
  Interventions: Behavioral: In-Person weight loss
- FIT weight loss (Experimental): Intervention materials will be provided and mailed weekly to participants. Participants will be provided with the BodyMedia® FIT System that includes a wearable device to monitor physical activity and energy expenditure, a display device to provide feedback on achievement of energy expenditure and physical activity goals, and web-based software to assist with self-monitoring of dietary intake and to provide feedback on goal achievement. Participants will attend one introductory session in which a tutorial of the components of the enhanced FIT System will be provided. Participants will receive a one-hour lesson on basic guidelines of the weight loss intervention. Once per month participants will receive a scheduled 10 minute intervention telephone call with the intervention staff.
  Interventions: Behavioral: FIT weight loss
- FIT-BT weight loss (Experimental): Participants will be provided with intervention materials that are mailed weekly to them. Participants will be provided with the enhanced BodyMedia® FIT System that includes a wearable device with Bluetooth® technology to allow participants to receive real-time feedback on calories expended and physical activity on their smart phone. This also supports self-monitoring of dietary behaviors and body weight. Participants will attend one introductory session in which a tutorial of the components of the enhanced FIT System will be provided. Participants will also receive a one-hour lesson on basic guidelines of the weight loss intervention. Once per month participants will receive a scheduled 10 minute intervention telephone call with the intervention staff.
  Interventions: Behavioral: FIT-BT weight loss

INTERVENTIONS:
Behavioral: In-Person weight loss — Participants will attend weekly group intervention meetings. These sessions will address barriers associated with altering physical activity participation and dietary intake. Group discussions will be facilitated by the interventionist and interactive participation will be encouraged. Participants will be provided with written materials at each meeting to supplement group discussions. Paper diaries will be provided each week to assist participants with self-monitoring of calorie and fat consumption, and physical activity minutes and intensity. Participants will return the diary to the intervention staff each week for review and constructive feedback.
  Arms: In-Person weight loss
Behavioral: FIT weight loss — Intervention materials will be provided and mailed weekly to participants. Participants will be provided with the BodyMedia® FIT System that includes a wearable device to monitor physical activity and energy expenditure, a display device to provide feedback on achievement of energy expenditure and physical activity goals, and web-based software to assist with self-monitoring of dietary intake and to provide feedback on goal achievement. Participants will attend one introductory session in which a tutorial of the components of the enhanced FIT System will be provided. Participants will receive a one-hour lesson on basic guidelines of the weight loss intervention. Once per month participants will receive a scheduled 10 minute intervention telephone call with the intervention staff.
  Arms: FIT weight loss
Behavioral: FIT-BT weight loss — Participants will be provided with intervention materials that are mailed weekly to them. Participants will be provided with the enhanced BodyMedia® FIT System that includes a wearable device with Bluetooth® technology to allow participants to receive real-time feedback on calories expended and physical activity on their smart phone. This also supports self-monitoring of dietary behaviors and body weight. Participants will attend one introductory session in which a tutorial of the components of the enhanced FIT System will be provided. Participants will also receive a one-hour lesson on basic guidelines of the weight loss intervention. Once per month participants will receive a scheduled 10 minute intervention telephone call with the intervention staff.
  Arms: FIT-BT weight loss

SUMMARY:
The purpose of this study is to examine the effect of an enhanced technology-based system, that involves a wearable device to measure calories burned combined with a website, in comparison to previous versions of similar technology and a standard behavioral weight loss on body weight across 6 months in obese adults.

DETAILED DESCRIPTION:
The primary aim of this study is to compare changes in body weight between an in-person behavioral weight loss program, a technology-based system, and an enhanced version of a technology-based system during a 6 month behavioral weight loss intervention in obese adults. Additional aims will compare changes in body composition, physical activity, dietary intake, and the frequency of self-monitoring of weight loss behaviors between the 3 groups. A total of 84 sedentary, healthy obese adults (BMI: 35.0-45.0 kg/m2) between the ages of 21-55 will be recruited to participate. Assessments will be conducted at 0, 3, and 6 months and will include measurements of height, weight, body composition, blood pressure, physical activity, dietary intake, and eating behaviors. This is a randomized controlled trial in which participants will be randomized after the completion of assessments to one of three groups: standard behavioral weight loss (SBWL), BodyMedia® FIT System (FIT), and BodyMedia® FIT System with Bluetooth® enhancements (FIT-BT). Subjects in SBWL will participate in a behavioral weight loss intervention which includes weekly group sessions throughout the 6 month program. FIT and FIT-BT will not attend weekly group sessions, but will have identical intervention materials mailed each week. FIT will receive the BodyMedia® FIT System, and FIT-BT will receive the BodyMedia® FIT System with Bluetooth® enhancements to use throughout the 6 month program. FIT and FIT-BT will receive a telephone intervention call 1x per month.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years of age
* Body mass index (BMI) between 35.0-45.0 kg/m2

Exclusion Criteria:

* Reports not having access to a computer, access to the Internet, or the availability to download software onto a computer.
* Reports not having a smart phone device that is compatible with the BodyMedia® FIT Bluetooth® System that will be examined in this study.
* Has a physical limitation that would prevent engaging in physical activity.
* Participates in structured aerobic exercise for ≥ 60 minutes per week over the prior ≥ 3 months.
* Reports being treated for a current medical condition that could affect body weight. These may include the following: cancer; diabetes mellitus; hyperthyroidism; inadequately controlled hypothyroidism; chronic renal insufficiency; chronic liver disease; gastrointestinal disorders including ulcerative colitis, Crohn's disease, or malabsorption syndromes, etc.
* Reports current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of increase risk of an acute cardiovascular event, coronary artery bypass grafting or angioplasty, prior myocardial infarction, and conditions requiring anticoagulation therapy (i.e. deep vein thrombosis).
* Has a resting systolic blood pressure ≥ 150 mmHg or resting diastolic blood pressure of ≥ 100 mmHg or taking medications to control blood pressure.
* Being treated for any psychological issues (i.e., depression, bipolar disorder, etc) or taking psychotropic medications within the previous 12 months.
* Taking prescription or over-the-counter medications that affect body weight and metabolism.
* Has lost > 5% of current body weight in the past 3 months and maintained this weight loss at the time of recruitment for this study.
* Currently participating in an exercise or weight control study, had participated in an exercise or weight control study within the previous 6 months, or a current participant in a commercial weight reduction program.
* Has undergone bariatric surgery (e.g., gastric bypass, lap-band) for weight loss.
* Currently being treated for an eating disorder.
* Currently pregnant, pregnant in the last 6 months, breast feeding in the last 3 months, lactating, to planning on becoming pregnant in the next 3 months.
* Planning on relocating outside of the greater Pittsburgh area within the next 6 months.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Change in body composition | Baseline, 3 months, and 6 months
Change in moderate-to-vigorous intensity physical activity | Baseline, 3 months, and 6 months
Change in dietary intake | Baseline, 3 months, and 6 months
Completion of self-monitoring of eating behavior | Baseline to 6 months
  The frequency that participants engaged in the self-monitoring of eating behavior as measured by either completion of an eating diary or the use of the BodyMedia Fit system software.
Frequency of self-monitoring of physical activity behavior | Baseline to 6 months
  The frequency that participants engaged in the self-monitoring of physical activity as measured by either completion of an exercise diary or the use of the BodyMedia Fit system.

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, PhD, Principal Investigator — University of Pittsburgh; Renee J Rogers, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States